CLINICAL TRIAL: NCT05821790
Title: Role of the Tumor Microenvironment in Aggressive Meningiomas
Acronym: MEME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Paris Brain Institute (Unknown); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230289
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Meningioma
Keywords: meningioma; meningeal lymphatic vessels; NF2; meningeal micro-environment; immune cells; neurosurgery
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients treated for meningioma: Samples required for the study will be obtained from surgical waste of patients who underwent meningioma resection.
  Interventions: Other: Surgical waste and Data collect

INTERVENTIONS:
Other: Surgical waste and Data collect — Samples required for the study will be obtained from surgical waste of patients who underwent meningioma resection. Data necessary for the study will be collected from the patient's medical records, MRI examinations, and data specific to the characteristics of the surgical waste.

SUMMARY:
Meningiomas are the most common primary tumors of the central nervous system in adults. High-grade forms have a high frequency of neurofibromatosis 2 (NF2) mutations and represent 25% of meningiomas, with multiple recurrences associated with morbidity and reduced survival without medical options, including immunotherapy. The meninges play a key role in neuro-immune communication through the diversity of their immune cells and the presence of meningeal lymphatic vessels (MLV). Recent data, including from our team, shows frequent infiltration of lymphocytes and myeloid cells specific to benign meningiomas. Our hypothesis is that the immune microenvironment composed of meningeal immune cells and MLVs regulates the malignant histological progression of NF2-mutated meningiomas and their immune surveillance evasion behavior This study aims to characterize the different cellular populations of the meningioma microenvironment. We will describe the exact participation of immune and vascular cell populations in the initiation and progression of meningioma, using MRI imaging and surgical biopsies of the dura mater and meningioma in patients undergoing neurosurgery for meningioma resection.

DETAILED DESCRIPTION:
The objective of this study is to characterize the different cellular populations of the microenvironment of meningioma, particularly the immune and vascular cell populations, in order to better understand their role in the initiation and progression of this tumor. For this purpose, we will use MRI imaging and surgical biopsies of the dura mater and meningioma to characterize cellular phenotypes and their interactions in the tissue microenvironment. The research will be conducted on a cohort of patients treated for meningioma in neurosurgery services. Samples required for the study will be obtained from surgical waste of patients who underwent meningioma resection. Data necessary for the study will be collected from the patient's medical records, MRI examinations, and data specific to the characteristics of the surgical waste. Prospective patients will be informed of the study through an information note. Patients who do not object to their participation will undergo neurosurgery intervention in accordance with the usual service protocol. During the intervention, surgical waste will be produced, including the meningioma and adjacent dura mater, which will be collected under the responsibility of the neuro-pathologist who will also take fragments for routine diagnostic histological analysis. We will then perform a targeted mutational analysis associated with neuropathological evaluation of the tumor grade in order to select 10 cases of grade I meningioma and 10 cases of grade II and III meningioma carrying the NF2 mutation. An in-depth analysis will then be carried out on these samples using 10x Genomic's single-cell RNA sequencing (scRNA-seq) technology. This analysis will help to understand the tumor's heterogeneity and establish the phenotype and differentiation trajectory of tumor cells, dura mater cells, and associated immune cells. In addition to RNA analysis, the expression of genetic signatures will be validated by RNAscope tests, while Hyperion imaging will allow visualization of the interrelationships between different types of cells and their spatial distribution. The iDISCO+ immunolabeling combined with three-dimensional fluorescence microscopy imaging will enable visualization of specific protein expression profiles of meningioma and dura mater cell types in 3D. Once the analyses are complete, meningioma and dura mater samples will be destroyed. Preoperative MRI images will also be retrieved and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent surgery for the resection of a meningioma.
2. Patients with meningiomas located at the convexity and parasagittal regions.
3. Patients aged 18 years or older.
4. Patients who were informed of the study and did not express opposition to their participation.

Exclusion Criteria:

* Individuals under legal protection (guardianship, trusteeship) safeguarded by justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery for the resection of a meningioma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Cellular phenotypes and their interactions in the tissue microenvironment | one day
  Characterized by combining different techniques and analysis systems (RNA-seq, RNAScope, Hyperion, Hyperion immunostaining) using samples from various grades of meningiomas and associated dura mater

SECONDARY OUTCOMES:
Expressed genes in meningioma | one day
  Differential expression and gene ontology of expressed genes in meningioma cells, dura mater cells, and associated immune cells, obtained through scRNA-seq and RNAscope analyses using samples from various grades of meningiomas and dura mater
cell types and spatial distribution | One day
  The cell types and their spatial distribution in meningiomas and associated dura mater characterized by the Hyperion cellular imaging system
Visualization of interrelations in the spatial context | One day
  Using the Hyperion cellular imaging system
3D protein expression | One day
  Specific 3D protein expression profiles of cell type in meningiomas and associated dura mater obtained through iDISCO+ immunolabeling combined with fluorescence microscopy imaging
Three-dimensional reconstruction | One day
  Three-dimensional reconstruction of the lymphatic vessels and their cervical lymph nodes associated with pre-surgery MRI data.

CONTACTS AND LOCATIONS:
Overall Officials: Michel KALAMARIDES, MD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No